CLINICAL TRIAL: NCT03670875
Title: Non-Pharmacologic Alternatives for the Treatment of Childhood Obesity in Mexico
Brief Title: Non-Pharmacologic Alternatives for Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Fernando Guerrero Romero MD, Head of the research unit, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2016-785-103
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Obesity in Childhood
Keywords: Children, obesity, agave-inulin, curcumin, O3FA
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Study groups. Agave inulin: 2.3 g twice a day by mouth during 3 months plus recommendations to decrease calories intake an do exercise.
  Curcumin: 600 mg (turmeric 600 + black pepper 5 mg) by mouth daily during 3 months plus recommendations to decrease calories intake an do exercise.
  Omega-3 fatty acids 600 mg (eicosapentaenoic acid 360; docosahexaenoic acid 240) Three times a day by mouth during 3 months plus recommendations to decrease calories intake an do exercise.
  Control group with no intervention. Recommendations to decrease calories intake an do exercise.
  Dietary recommendations to ingest 1600 calories per day Exercise: 30 minutes each day, al least 5 days a week (caloric consumption 150-200 kcal per day)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Agave inulin (Experimental): Agave inulin 2.3 g, by mouth, every 12 hours for 3 months. Plus recommendations to decrease calories intake an do exercise.
  Interventions: Dietary Supplement: Agave inulin
- Curcumin (Experimental): Curcumin 600 mg (turmeric 600 + black pepper 5 mg) by mouth, daily for 3 months. Plus recommendations to decrease calories intake an do exercise.
  Interventions: Dietary Supplement: Curcumin
- Omega 3 Fatty Acids (Experimental): O3FA 600 mg (eicosapentaenoic acid 360; docosahexaenoic acid 240) Three times a day by mouth, every 8 hours for 3 months. Plus recommendations to decrease calories intake an do exercise.
  Interventions: Dietary Supplement: O3FA
- Control (Other): Recommendations to decrease calories intake an do exercise.
  Interventions: Behavioral: Control

INTERVENTIONS:
Dietary Supplement: Agave inulin — Will be provided in dehydrated apple cubes
  Arms: Agave inulin
Dietary Supplement: Curcumin — Will be provided in capsules
  Other Names: Turmeric
  Arms: Curcumin
Dietary Supplement: O3FA — Will be provided in capsules
  Arms: Omega 3 Fatty Acids
Behavioral: Control — Dietary recommendations to ingest 1600 calories per day. Exercise: 30 minutes each day, al least 5 days a week (caloric consumption 150-200 kcal per day)
  Arms: Control

SUMMARY:
Childhood obesity is a global health issue. Mexico has been considered as the country with the higher number of children with obesity. There are not approved drugs to support diet and exercise as the first step to lose weight. Animal models and clinical trials in adults have provided evidence about safety and efficacy of interventions such as: prebiotics, curcumin, and omega- 3 fatty acids. The hypothesis of this study is: that non-pharmacological alternatives could support diet and exercise to decrease the weight of children with obesity.

DETAILED DESCRIPTION:
The aim of this study is to determinate the efficacy and safety of agave inulin, curcumin, and omega-3 fatty acids (O3FA) to decrease the weight of children with obesity.

Design. Randomized controlled clinical trial (RCT) with four study groups: agave inulin, curcumin, omega-3 fatty acids and a control group. All groups will receive instructions to decrease calories intake and do exercise.

Children sent to the unit with a presumptive diagnosis of obesity will be considered as candidates to the RCT. Children accomplishing with inclusion/exclusion criteria will be randomized to one of the study groups.

Sample size was calculated using a statistical power of 80%, alpha value of 0.05. A 15 % of difference, in the mean of weight reduction, between control group and intervention groups was considered. The estimated sample size was 75 subjects for each group.

Weight, height, BMI, blood pressure, abdominal circumference and body fat percentage will be measured in months 0, 1, 2, and 3. In months 0 and 3 a fasting venous blood sample will be drawn to perform the following test: glucose, insulin, lipid profile and C- Reactive protein, aspartate aminotransferase (AST) and alanine aminotransferase (ALT). Anthropometric measures, food intake recommendation and diaries of food consume will be performed by trained nutritionists. Recommendation about type of exercise and estimation of calories consumed will be performed by a physical education teacher.

The statistical analysis will performed by one to the investigators blinded to treatment groups. Numerical values will be expressed as mean ± standard deviation. Categorical variables will be expressed as proportions. The analysis will be preformed according with CONSORT group recommendations Differences between the groups were estimated using one-way ANOVA with Bonferroni post-hoc test for numerical parameters and χ 2 test for categorical variables. Intragroup differences will be assessed by paired Student t test (Mann-Whitney U test for skewed data). Statistical significance will be considered as a p value <0.05 and 95% confidence interval (CI). Statistical Package for the Social Sciences will be used for the analysis

ELIGIBILITY:
Inclusion Criteria:

* Gender: Boys and Girls
* Diagnosis of obesity (percentile ≥ 95% according to The Centers for Disease Control and Prevention growth charts)
* Informed consent of parents
* Informed assent of the participant

Exclusion criteria:

* Diabetes
* Thyroid disease
* Renal disease
* Hepatic disease
* Neoplasia disease
* Chronic gastrointestinal conditions
* Consume of prebiotics or probiotics
* Consume of prebiotics or food supplements
* Use of anti-inflammatory drugs.
* Recent use of antibiotics (30 days)

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Loosing weight | Three months
  Weight lost between basal and third month visits. Determined by a digital scale

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Guerrero, PhD, Principal Investigator — Instituto Mexicano del Seguro Social; Gerardo Martinez, PhD, Study Director — Instituto Mexicano del Seguro Social; Luis E Simental, PhD, Study Chair — Instituto Mexicano del Seguro Social; Claudia I Gamboa, PhD, Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Biomedical Research Unit. IMSS. Durango, Durango, Durango, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gluckman P, Nishtar S, Armstrong T. Ending childhood obesity: a multidimensional challenge. Lancet. 2015 Mar 21;385(9973):1048-50. doi: 10.1016/S0140-6736(15)60509-8. No abstract available. PMID 25797547
- [Background] Siro I, Kapolna E, Kapolna B, Lugasi A. Functional food. Product development, marketing and consumer acceptance--a review. Appetite. 2008 Nov;51(3):456-67. doi: 10.1016/j.appet.2008.05.060. Epub 2008 Jun 4. PMID 18582508
- [Background] Tomaschunas M, Zorb R, Fischer J, Kohn E, Hinrichs J, Busch-Stockfisch M. Changes in sensory properties and consumer acceptance of reduced fat pork Lyon-style and liver sausages containing inulin and citrus fiber as fat replacers. Meat Sci. 2013 Nov;95(3):629-40. doi: 10.1016/j.meatsci.2013.06.002. Epub 2013 Jun 10. PMID 23811098
- [Background] Mancilla-Margalli NA, Lopez MG. Water-soluble carbohydrates and fructan structure patterns from Agave and Dasylirion species. J Agric Food Chem. 2006 Oct 4;54(20):7832-9. doi: 10.1021/jf060354v. PMID 17002459
- [Background] González-Herrera SM, Rutiaga-Quiñones OM, Aguilar CN, et al. Dehydrated Apple matrix supplemented with agave fructans, inulin and oligofructose. LWT Food Science and Technology. 2016;65:1059-1065.
- [Background] Lopez-Velazquez G, Diaz-Garcia L, Anzo A, Parra-Ortiz M, Llamosas-Gallardo B, Ortiz-Hernandez AA, Mancilla-Ramirez J, Cruz-Rubio JM, Gutierrez-Castrellon P. Safety of a dual potential prebiotic system from Mexican agave "Metlin(R) and Metlos(R)", incorporated to an infant formula for term newborn babies: a randomized controlled trial. Rev Invest Clin. 2013 Nov-Dec;65(6):483-90. PMID 24687355
- [Background] Wang SL, Li Y, Wen Y, Chen YF, Na LX, Li ST, Sun CH. Curcumin, a potential inhibitor of up-regulation of TNF-alpha and IL-6 induced by palmitate in 3T3-L1 adipocytes through NF-kappaB and JNK pathway. Biomed Environ Sci. 2009 Feb;22(1):32-9. doi: 10.1016/S0895-3988(09)60019-2. PMID 19462685
- [Background] Sahebkar A. Why it is necessary to translate curcumin into clinical practice for the prevention and treatment of metabolic syndrome? Biofactors. 2013 Mar-Apr;39(2):197-208. doi: 10.1002/biof.1062. Epub 2012 Dec 13. PMID 23239418
- [Background] Ramirez-Bosca A, Soler A, Carrion MA, Diaz-Alperi J, Bernd A, Quintanilla C, Quintanilla Almagro E, Miquel J. An hydroalcoholic extract of curcuma longa lowers the apo B/apo A ratio. Implications for atherogenesis prevention. Mech Ageing Dev. 2000 Oct 20;119(1-2):41-7. doi: 10.1016/s0047-6374(00)00169-x. PMID 11040400
- [Background] Nagwa I, Ragab S, Baky A, et al. Effect of Oral Curcumin Administration on Insulin Resistance, Serum Resistin and Fetuin-A in Obese Children: Randomized Placebo- Controlled study. Reser J of Pharm, Biol and Chem Sci 2014 5:887-96
- [Background] Suskind DL, Wahbeh G, Burpee T, Cohen M, Christie D, Weber W. Tolerability of curcumin in pediatric inflammatory bowel disease: a forced-dose titration study. J Pediatr Gastroenterol Nutr. 2013 Mar;56(3):277-9. doi: 10.1097/MPG.0b013e318276977d. PMID 23059643
- [Background] Huang XF, Xin X, McLennan P, Storlien L. Role of fat amount and type in ameliorating diet-induced obesity: insights at the level of hypothalamic arcuate nucleus leptin receptor, neuropeptide Y and pro-opiomelanocortin mRNA expression. Diabetes Obes Metab. 2004 Jan;6(1):35-44. doi: 10.1111/j.1463-1326.2004.00312.x. PMID 14686961
- [Background] Couet C, Delarue J, Ritz P, Antoine JM, Lamisse F. Effect of dietary fish oil on body fat mass and basal fat oxidation in healthy adults. Int J Obes Relat Metab Disord. 1997 Aug;21(8):637-43. doi: 10.1038/sj.ijo.0800451. PMID 15481762
- [Background] Juarez-Lopez C, Klunder-Klunder M, Madrigal-Azcarate A, Flores-Huerta S. Omega-3 polyunsaturated fatty acids reduce insulin resistance and triglycerides in obese children and adolescents. Pediatr Diabetes. 2013 Aug;14(5):377-83. doi: 10.1111/pedi.12024. Epub 2013 Feb 25. PMID 23438101
- [Background] Parra D, Ramel A, Bandarra N, Kiely M, Martinez JA, Thorsdottir I. A diet rich in long chain omega-3 fatty acids modulates satiety in overweight and obese volunteers during weight loss. Appetite. 2008 Nov;51(3):676-80. doi: 10.1016/j.appet.2008.06.003. Epub 2008 Jun 14. PMID 18602429